CLINICAL TRIAL: NCT03533491
Title: Mindfulness Mobile App to Reduce Adolescent Substance Use
Brief Title: The Rewire Study (Mindfulness Mobile App to Reduce Adolescent Substance Use)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Research Behavioral Intervention Strategies, Inc. (Industry)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DA043288-01; 1R43DA043288-01 (NIH)
Record Dates: First submitted 2018-04-17; First posted 2018-05-23 (Actual); Results first posted 2024-11-13 (Actual); Last update posted 2024-11-13 (Actual); Status verified 2024-10

CONDITIONS: Adolescent Substance Use

STUDY DESIGN:
Intervention Model Description: All 60 teens in The Rewire Study will complete the first 4 modules of the Rewire app.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- App Evaluation (Experimental): All 60 teens in The Rewire Study will complete the first 4 modules of the Rewire app. Prior to using the app, they will complete a baseline assessment. Follow up surveys will be completed at 2 weeks and 8 weeks post-baseline.
  Interventions: Behavioral: Rewire App

INTERVENTIONS:
Behavioral: Rewire App — A prototype Rewire app will be designed and created; the first four modules will be evaluated by 60 high-risk adolescents. The teens are asked to complete each module and spend a few minutes each day for two weeks using the practice exercises.

SUMMARY:
The current proposal is aimed at developing a substance use cessation app (Rewire) for high risk adolescents who are involved in the juvenile justice system. The Rewire app will be based on the primary substance use cessation components tested in our previous work with juvenile justice-involved adolescents and on intervention components shown to be central to smoking cessation.

DETAILED DESCRIPTION:
The Rewire Study will recruit 60 youth (30 boys and 30 girls) who have had contact with the Department of Youth Services in the last year. Consent will be obtained from parents or guardians for the youths' participation. The participating teens will come to Oregon Research Institute for a baseline assessment. During this visit, the teens will complete an assent form and spend 20-30 minutes completing an online survey with an assessor; topics covered in the survey include emotion regulation and drug and alcohol use. Teens will have the app loaded onto their phones and be provided with instructions for its use during this visit. Participants are asked to use the app over the next 2 weeks, completing 4 modules and spending 5-10 minutes each day answering questions about recent emotions and substance use. Teens will be contacted via email for follow up assessments at 8 weeks post-baseline. These emails will contain links to the follow-up surveys which also ask about emotion regulation and drug and alcohol use; surveys should take 20-30 minutes to complete.

ELIGIBILITY:
Inclusion Criteria:

* ages 13 to 18
* involved with Juvenile Justice system
* documented substance use
* English-speaking
* living in the community

Exclusion Criteria:

* non English-speaking
* living in treatment or detention facility

Ages: 13 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Actual)
Dates: Start 2018-03-30 (Actual); Primary Completion 2018-08-30 (Actual); Study Completion 2018-10-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dana K Smith, Ph.D., Principal Investigator — Oregon Research Institute
Locations (1):
- Oregon Research Behavioral Intervention Strategies, Inc./Oregon Research Institute, Eugene, Oregon, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | App Evaluation
Started | 60
Completed | 58
Not Completed | 2
Not completed — Lost to Follow-up | 2

BASELINE CHARACTERISTICS:
Arm/Group | App Evaluation
Number analyzed (Participants) | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 15.57 (1.42)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30
  Male | 30
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 38
  More than one race | 6
  Unknown or Not Reported | 13

OUTCOME MEASURES:

1. Primary Outcome: Adolescent Use of Cigarettes
Description: Proportion of participants that use cigarettes as measured by Youth Substances Interview
Time Frame: Baseline (pretest), 8 weeks (posttest)
Measure: Mean (Standard Deviation); unit: proportion of participants
Arm/Group | App Evaluation
Number analyzed (Participants) | 58
proportion of participants
  Pretest | 0.19 (0.40)
  Posttest | 0.12 (0.33)
Statistical Analysis 1: Comparison: App Evaluation; Test type: Equivalence — A test of the null hypothesis that the proportion of participants from pretest to posttest change is equal to zero; p = .044, t-test, 2 sided; Proportion Difference = .070, Standard Error of Mean .044 — A paired t-test that evaluates whether significant pretest to posttest change in the proportion of users is different from zero

2. Primary Outcome: Adolescent Use of E-cigarettes
Description: Proportion of participants that use e-cigarette use as measured by Youth Substances Interview
Time Frame: Baseline (pretest), 8 weeks (posttest)
Measure: Mean (Standard Deviation); unit: proportion of participants
Arm/Group | App Evaluation
Number analyzed (Participants) | 58
proportion of participants
  Pretest | 0.32 (0.47)
  Posttest | 0.28 (0.45)
Statistical Analysis 1: Comparison: App Evaluation; Test type: Equivalence — A test of the null hypothesis that the proportion who use from pretest to posttest is equal to zero; p = .532, t-test, 2 sided; A paired t-test that evaluates whether the proportion who use from pretest to posttest change is different from zero; Proportion Difference = .035, Standard Error of Mean .056

3. Primary Outcome: Adolescent Use of Alcohol
Description: Proportion of participants that use alcohol use as measured by Youth Substances Interview
Time Frame: Baseline (pretest), 8 weeks (posttest)
Measure: Mean (Standard Deviation); unit: proportion of participants
Arm/Group | App Evaluation
Number analyzed (Participants) | 58
proportion of participants
  Pretest | 0.39 (0.49)
  Posttest | 0.44 (0.50)
Statistical Analysis 1: Comparison: App Evaluation; Test type: Equivalence — A test of the null hypothesis that the proportion of participants who use from pretest to posttest is equal to zero; p = .370, t-test, 2 sided; A paired t-test that evaluates whether significant pretest to posttest change is different from zero; Proportion Difference = -.053, Standard Error of Mean .058

4. Primary Outcome: Adolescent Use of Marijuana
Description: Proportion of participants that use marijuana use as measured by Youth Substances Interview
Time Frame: Baseline (pretest), 8 weeks (posttest)
Measure: Mean (Standard Deviation); unit: proportion of participants
Arm/Group | App Evaluation
Number analyzed (Participants) | 58
proportion of participants
  Pretest | 0.54 (0.50)
  Posttest | 0.40 (0.49)
Statistical Analysis 1: Comparison: App Evaluation; Test type: Equivalence — A test of the null hypothesis that the proportion of participants that use from pretest to posttest is equal to zero; p = .020, t-test, 2 sided; A paired t-test that evaluates whether proportion who use from pretest to posttest is different from zero; Proportion Difference = .140, Standard Error of Mean 0.06

5. Secondary Outcome: Changes in Adolescent Mindfulness Practices - Observe Subscale
Description: Mindfulness is measured using the Five Facet Mindfulness Questionnaire. Mindfulness (Baer et al. 2006) was assessed with a 5-point response option (1 = never or very rarely true, 5 = every often or always true) and mean scores were computed for each subscale. A higher score indicates greater levels of mindfulness. Subscales include observing (8 items), describing (8 items), acting with awareness (8 items), non-judging of inner experience (8 items), and non-reactivity to inner experience (7 items).
Time Frame: Baseline (pretest), 8 weeks (posttest)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | App Evaluation
Number analyzed (Participants) | 58
units on a scale
  Pretest | 3.08 (0.75)
  Posttest | 3.05 (0.87)
Statistical Analysis 1: Comparison: App Evaluation; Test type: Equivalence — A test of the null hypothesis that the pretest to posttest change is equal to zero; p = .773, t-test, 2 sided; A paired t-test that evaluates whether significant pretest to posttest change is different from zero; Mean Difference (Final Values) = .031, Standard Error of Mean .108

6. Secondary Outcome: Changes in Adolescent Mindfulness Practices - Describing Subscale
Description: as for outcome 5
Time Frame: Baseline (pretest) and 8-weeks (posttest)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | App Evaluation
Number analyzed (Participants) | 58
units on a scale
  Pretest | 3.29 (0.68)
  Posttest | 3.28 (0.73)
Statistical Analysis 1: Comparison: App Evaluation; Test type: Equivalence — A test of the null hypothesis that the pretest to posttest change is equal to zero; p = .978, t-test, 2 sided; A paired t-test that evaluates whether significant pretest to posttest change is different from zero; Mean Difference (Final Values) = .002, Standard Error of Mean .080

7. Secondary Outcome: Change in Adolescent Mindfulness Practices - Acting With Awareness Subscale
Description: as for outcome 5
Time Frame: Baseline (pretest) and 8-week (posttest)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | App Evaluation
Number analyzed (Participants) | 58
units on a scale
  Pretest | 2.89 (0.48)
  Posttest | 2.86 (0.57)
Statistical Analysis 1: Comparison: App Evaluation; Test type: Equivalence — A test of the null hypothesis that the pretest to posttest change is equal to zero; p = .745, t-test, 2 sided; A paired t-test that evaluates whether significant pretest to posttest change is different from zero; Mean Difference (Final Values) = .029, Standard Error of Mean .089

8. Secondary Outcome: Change in Adolescent Mindfulness Practices - Non-judging of Inner Experiences Subscale
Description: as for outcome 5
Time Frame: Baseline (pretest) and 8-weeks (posttest)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | App Evaluation
Number analyzed (Participants) | 58
units on a scale
  Pretest | 3.52 (0.81)
  Posttest | 3.37 (0.79)
Statistical Analysis 1: Comparison: App Evaluation; Test type: Equivalence — A test of the null hypothesis that the pretest to posttest change is equal to zero; p = .132, t-test, 2 sided; A paired t-test that evaluates whether significant pretest to posttest change is different from zero; Mean Difference (Final Values) = -.154, Standard Error of Mean .101

9. Secondary Outcome: Change in Adolescent Mindfulness Practices - Non-reactivity to Inner Experience Subscale
Description: as for outcome 5
Time Frame: Baseline (pretest) and 8-week (posttest)
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | App Evaluation
Number analyzed (Participants) | 58
units on a scale
  Pretest | 2.97 (0.65)
  Posttest | 2.91 (0.81)
Statistical Analysis 1: Comparison: App Evaluation; Test type: Equivalence — A test of the null hypothesis that the pretest to posttest change is equal to zero; p = .551, t-test, 2 sided; A paired t-test that evaluates whether significant pretest to posttest change is different from zero; Mean Difference (Final Values) = .066, Standard Error of Mean .111

10. Secondary Outcome: Changes in Emotion Regulation - Non-acceptance of Emotional Response Subscale
Description: Emotion Regulation is measured with the Difficulties in Emotion Regulation Scale. Emotional regulation (Gratz and Roemer, 2004) was assessed with a 5-point response option (1 = almost never, 5 = almost always) and mean scores were computed for each subscale. A higher score indicates greater levels of emotional regulation. Subscales include non-acceptance of emotional response (6 items), difficulties engaging in goals (5 items), impulse control difficulties (6 items), lack of emotional awareness (6 items), limited access to emotion regulation strategies (8 items), and lack of emotional clarity (6 items).
Time Frame: Baseline (pretest), 8 weeks (posttest)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | App Evaluation
Number analyzed (Participants) | 58
units on a scale
  Pretest | 1.93 (0.86)
  Posttest | 2.09 (1.05)
Statistical Analysis 1: Comparison: App Evaluation; Test type: Equivalence — A test of the null hypothesis that the pretest to posttest change is equal to zero; p = .255, t-test, 2 sided; A paired t-test that evaluates whether significant pretest to posttest change is different from zero; Mean Difference (Final Values) = -.158, Standard Error of Mean .255

11. Secondary Outcome: Changes in Emotional Regulation - Difficulties Engaging in Goals Subscale
Description: as for outcome 10
Time Frame: Baseline (pretest) and 8-weeks (posttest)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | App Evaluation
Number analyzed (Participants) | 58
units on a scale
  Pretest | 2.83 (1.02)
  Posttest | 2.69 (1.09)
Statistical Analysis 1: Comparison: App Evaluation; Test type: Equivalence — A test of the null hypothesis that the pretest to posttest change is equal to zero; A paired t-test that evaluates whether significant pretest to posttest change is different from zero; Mean Difference (Final Values) = .139, Standard Error of Mean .142

12. Secondary Outcome: Changes in Emotional Regulation - Impulse Control Difficulties Subscale
Description: as for outcome 10
Time Frame: Baseline (pretest) and 8-weeks (posttest)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | App Evaluation
Number analyzed (Participants) | 58
units on a scale
  Pretest | 1.86 (0.92)
  Posttest | 1.98 (0.87)
Statistical Analysis 1: Comparison: App Evaluation; Test type: Equivalence — A test of the null hypothesis that the pretest to posttest change is equal to zero; p = .198, t-test, 2 sided; Mean Difference (Final Values) = -.119, Standard Error of Mean .091

13. Secondary Outcome: Changes in Emotional Regulation - Lack of Emotional Awareness Subscale
Description: as for outcome 10
Time Frame: Baseline (pretest) and 8-weeks (Posttest)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | App Evaluation
Number analyzed (Participants) | 58
units on a scale
  Pretest | 2.79 (0.87)
  Posttest | 2.82 (0.96)
Statistical Analysis 1: Comparison: App Evaluation; Test type: Equivalence — A test of the null hypothesis that the pretest to posttest change is equal to zero; p = .770, t-test, 2 sided; A paired t-test that evaluates whether significant pretest to posttest change is different from zero; Mean Difference (Final Values) = -.035, Standard Error of Mean .121

14. Secondary Outcome: Changes in Emotional Regulation - Limited Access to Emotion Regulation Strategies Subscale
Description: as for outcome 10
Time Frame: Baseline (pretest) and 8-week (posttest)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | App Evaluation
Number analyzed (Participants) | 58
units on a scale
  Pretest | 2.22 (1.05)
  Posttest | 2.25 (1.03)
Statistical Analysis 1: Comparison: App Evaluation; Test type: Equivalence — A test of the null hypothesis that the pretest to posttest change is equal to zero; p = .834, t-test, 2 sided; A paired t-test that evaluates whether significant pretest to posttest change is different from zero; Mean Difference (Final Values) = -.029, Standard Error of Mean .137

15. Secondary Outcome: Changes in Emotional Regulation - Lack of Emotional Clarity
Description: as for outcome 10
Time Frame: Baseline (pretest) and 8-weeks (posttest)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | App Evaluation
Number analyzed (Participants) | 58
units on a scale
  Pretest | 2.22 (0.71)
  Posttest | 2.31 (0.77)
Statistical Analysis 1: Comparison: App Evaluation; Test type: Equivalence — A test of the null hypothesis that the pretest to posttest change is equal to zero; p = .175, t-test, 2 sided; A paired t-test that evaluates whether significant pretest to posttest change is different from zero; Mean Difference (Final Values) = -.096, Standard Error of Mean .070

ADVERSE EVENTS:
Time Frame: From enrollment in study through completion, an average of 8 weeks
Arm/Group | App Evaluation
All-Cause Mortality (participants affected / at risk) | 0/60
Serious Adverse Events (participants affected / at risk) | 0/60
Other Adverse Events (participants affected / at risk) | 0/60

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2017-04-17): https://cdn.clinicaltrials.gov/large-docs/91/NCT03533491/Prot_SAP_000.pdf
  • Informed Consent Form (2018-02-20): https://cdn.clinicaltrials.gov/large-docs/91/NCT03533491/ICF_001.pdf